CLINICAL TRIAL: NCT03268005
Title: Efficacy and Safety of Fast-acting Insulin Aspart Compared to NovoRapid® Both in Combination With Insulin Degludec With or Without Metformin in Adults With Type 2 Diabetes (Onset® 9)
Brief Title: Research Study Comparing a New Medicine "Fast-acting Insulin Aspart" to Another Already Available Medicine "NovoRapid"/"NovoLog" in People With Type 2 Diabetes
Acronym: onset 9
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN1218-4113; U1111-1180-0636 (Other: World Health Organization (WHO)); 2016-000878-38 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Results first posted 2020-03-12 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart; insulin degludec; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Faster aspart + insulin degludec with or without metformin (Experimental)
  Interventions: Drug: Faster-acting insulin aspart; Drug: Insulin degludec; Drug: Metformin
- NovoRapid/NovoLog + insulin degludec with or without metformin (Active Comparator)
  Interventions: Drug: Insulin aspart; Drug: Insulin degludec; Drug: Metformin

INTERVENTIONS:
Drug: Faster-acting insulin aspart — Faster aspart given subcutaneously (s.c., under the skin) once a day for 16 weeks. Dose individually adjusted.
  Arms: Faster aspart + insulin degludec with or without metformin
Drug: Insulin aspart — Insulin aspart given subcutaneously (s.c., under the skin) once a day for 16 weeks. Dose individually adjusted.
  Arms: NovoRapid/NovoLog + insulin degludec with or without metformin
Drug: Insulin degludec — Insulin degludec given subcutaneously (s.c., under the skin) once a day for 16 weeks. Dose individually adjusted.
Drug: Metformin — Only participants who took metformin before the study should take metformin tablets, same dose as before the study

SUMMARY:
The study compares 2 medicines for type 2 diabetes: fast-acting insulin aspart (a new medicine) and NovoRapid®/NovoLog® (a medicine doctors can already prescribe). Fast-acting insulin aspart will be tested to see how well it works and if it is safe. Participants will get either fast-acting insulin aspart or NovoRapid®/ NovoLog® - which treatment you get is decided by chance. Both medicines will be taken together with insulin degludec. Participants will need to take 1 injection 4 times every day (all insulins will be provided in pens). The study will last for about 8 months (34 weeks).

ELIGIBILITY:
Inclusion Criteria: - Male or female, age equal to or above 18 years at the time of signing informed consent. - Diagnosed with type 2 diabetes mellitus for 10 years or longer prior to screening (Visit 1). - Treated with a basal-bolus insulin regimen for 1 year or longer prior to the day of screening (Visit 1). A basal-bolus insulin regimen is defined as basal insulin once or twice daily and bolus insulin analogue taken with meals at least 3 times daily. Treatment with premixed insulin or soluble insulin combination is not considered a basal-bolus regimen. - Treated with or without oral antidiabetic drugs including extended release formulations. - HbA1c 7.0-10.0% (both inclusive) as assessed by central laboratory at screening (Visit 1). Exclusion Criteria: - Any of the following: myocardial infarction, stroke, hospitalization for unstable angina or transient ischaemic attack within the past 180 days prior to the day of screening (Visit 1). - Subjects presently classified as being in New York Heart Association (NYHA) Class IV. - Planned coronary, carotid or peripheral artery revascularisation known on the day of screening (Visit 1). - Treatment with injectable GLP-1 receptor agonists in a period of 90 days prior to screening (Visit 1). - Anticipated initiation or change in concomitant medications (for more than 14 consecutive days) known to affect weight or glucose metabolism (e.g. treatment with orlistat, thyroid hormones, or corticosteroids).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1264 (Actual)
Dates: Start 2017-09-19 (Actual); Primary Completion 2019-01-07 (Actual); Study Completion 2019-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (144):
- United States (59):
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Fullerton, California
  - Novo Nordisk Investigational Site, Lancaster, California
  - Novo Nordisk Investigational Site, Norco, California
  - Novo Nordisk Investigational Site, Sacramento, California
  - Novo Nordisk Investigational Site, Ventura, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Boynton Beach, Florida
  - Novo Nordisk Investigational Site, Bradenton, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Alpharetta, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Honolulu, Hawaii
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Peoria, Illinois
  - Novo Nordisk Investigational Site, Springfield, Illinois
  - Novo Nordisk Investigational Site, Valparaiso, Indiana
  - Novo Nordisk Investigational Site, West Des Moines, Iowa
  - Novo Nordisk Investigational Site, Topeka, Kansas
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Waltham, Massachusetts
  - Novo Nordisk Investigational Site, Worcester, Massachusetts
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Mentor, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Greenville, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Nashville, Tennessee
  - Novo Nordisk Investigational Site, Amarillo, Texas
  - Novo Nordisk Investigational Site, Austin, Texas
  - Novo Nordisk Investigational Site, Beaumont, Texas
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Longview, Texas
  - Novo Nordisk Investigational Site, Pearland, Texas
  - Novo Nordisk Investigational Site, Round Rock, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Bennington, Vermont
  - Novo Nordisk Investigational Site, South Burlington, Vermont
  - Novo Nordisk Investigational Site, Chesapeake, Virginia
  - Novo Nordisk Investigational Site, Winchester, Virginia
  - Novo Nordisk Investigational Site, Olympia, Washington
  - Novo Nordisk Investigational Site, Seattle, Washington
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Green Bay, Wisconsin
- Argentina (2):
  - Novo Nordisk Investigational Site, CABA
  - Novo Nordisk Investigational Site, Córdoba
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Kozloduy
  - Novo Nordisk Investigational Site, Razgrad
  - Novo Nordisk Investigational Site, Sofia
- Canada (11):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Victoria, British Columbia
  - Novo Nordisk Investigational Site, Halifax, Nova Scotia
  - Novo Nordisk Investigational Site, Barrie, Ontario
  - Novo Nordisk Investigational Site, Concord, Ontario
  - Novo Nordisk Investigational Site, Etobicoke, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Newmarket, Ontario
  - Novo Nordisk Investigational Site, Thunder Bay, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Montreal, Quebec
- Croatia (4):
  - Novo Nordisk Investigational Site, Karlovac
  - Novo Nordisk Investigational Site, Osijek
  - Novo Nordisk Investigational Site, Varaždin
  - Novo Nordisk Investigational Site, Zagreb
- Czechia (3):
  - Novo Nordisk Investigational Site, Hradec Králové
  - Novo Nordisk Investigational Site, Pilsen
  - Novo Nordisk Investigational Site, Trutnov
- Germany (7):
  - Novo Nordisk Investigational Site, Dresden
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Falkensee
  - Novo Nordisk Investigational Site, Lingen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Saint Ingbert-Oberwürzbach
  - Novo Nordisk Investigational Site, Schweinfurt
- Greece (4):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Ioannina
  - Novo Nordisk Investigational Site, Larissa
  - Novo Nordisk Investigational Site, Thessaloniki
- Italy (6):
  - Novo Nordisk Investigational Site, Catanzaro
  - Novo Nordisk Investigational Site, Chieti
  - Novo Nordisk Investigational Site, Cittadella (PD)
  - Novo Nordisk Investigational Site, Milano (MI)
  - Novo Nordisk Investigational Site, Olbia
  - Novo Nordisk Investigational Site, Palermo
- Poland (4):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Skorzewo
  - Novo Nordisk Investigational Site, Warsaw
  - Novo Nordisk Investigational Site, Wroclaw
- Novo Nordisk Investigational Site, Ponce, Puerto Rico
- Romania (5):
  - Novo Nordisk Investigational Site, Baia Mare, Maramureş
  - Novo Nordisk Investigational Site, Târgu Mureş, Mureș County
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Brasov
  - Novo Nordisk Investigational Site, Bucharest
- Russia (7):
  - Novo Nordisk Investigational Site, Arkhangelsk
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Tyumen
  - Novo Nordisk Investigational Site, Voronezh
- Serbia (5):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Kragujevac
  - Novo Nordisk Investigational Site, Niš
  - Novo Nordisk Investigational Site, Novi Sad
  - Novo Nordisk Investigational Site, Zaječar
- Slovakia (5):
  - Novo Nordisk Investigational Site, Košice
  - Novo Nordisk Investigational Site, Kysucké Nové Mesto
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Ľubochňa
  - Novo Nordisk Investigational Site, Žilina
- South Korea (5):
  - Novo Nordisk Investigational Site, Bucheon-si
  - Novo Nordisk Investigational Site, Daegu
  - Novo Nordisk Investigational Site, Seongnam-si
  - Novo Nordisk Investigational Site, Seoul
  - Novo Nordisk Investigational Site, Wŏnju
- Spain (7):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Alcobendas
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Girona
  - Novo Nordisk Investigational Site, Pozuelo de Alarcón
  - Novo Nordisk Investigational Site, Sabadell
  - Novo Nordisk Investigational Site, Seville
- Ukraine (6):
  - Novo Nordisk Investigational Site, Dnipro
  - Novo Nordisk Investigational Site, Kharkiv
  - Novo Nordisk Investigational Site, Kyiv
  - Novo Nordisk Investigational Site, Lviv
  - Novo Nordisk Investigational Site, Ternopil
  - Novo Nordisk Investigational Site, Vinnytsia

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com

REFERENCES:
- [Result] Lane WS, Favaro E, Rathor N, Jang HC, Kjaersgaard MIS, Oviedo A, Rose L, Senior P, Sesti G, Soto Gonzalez A, Franek E. A Randomized Trial Evaluating the Efficacy and Safety of Fast-Acting Insulin Aspart Compared With Insulin Aspart, Both in Combination With Insulin Degludec With or Without Metformin, in Adults With Type 2 Diabetes (ONSET 9). Diabetes Care. 2020 Aug;43(8):1710-1716. doi: 10.2337/dc19-2232. Epub 2020 Mar 24. PMID 32209647
- [Derived] Lane W, Favaro E, Jodar E, Kelkar P, Oviedo A, Sivarathinasami R, Senior PA, Sesti G, Franek E. Effective Overall Glycaemic Control with Fast-Acting Insulin Aspart Across Patients with Different Baseline Characteristics: A Post Hoc Analysis of the Onset 9 Trial. Diabetes Ther. 2022 Apr;13(4):761-774. doi: 10.1007/s13300-022-01213-3. Epub 2022 Mar 15. PMID 35290624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 165 sites in 17 countries as follows: Argentina-3, Bulgaria-4, Canada-10, Croatia-4, Czech Republic-4, Germany-6, Greece-8, Italy-4, Poland-10, Republic of Korea-6, Romania-6, Russia-8, Serbia-9, Slovakia-5, Spain-8, Ukraine-6 and United States (US)-62. Two sites in the US screened but didn't randomise any subject.
Pre-assignment Details: There was a 12-week run-in period primarily for optimisation of the basal insulin and reinforcement of subject training in trial procedures, diabetes education and dietary training. Out of the 1264 participants enrolled in the study, 173 were run-in failures and 1091 were randomised.
Groups:
- Faster Aspart: Participants received Faster aspart along with insulin degludec (basal-bolus regimen) with or without metformin for 16 weeks. Before the treatment period was a 12-week run-in period in which the investigator optimised basal insulin dose. Insulin degludec dose was adjusted weekly by the investigator in the run-in period based on the mean of three pre-breakfast SMPG values measured on the last two days prior to and on the day of contact. If one of the SMPG values were below target (< 4.0 mmol/L or 71 mg/dL) then the insulin degludec dose was adjusted according to the titration guideline specified in the protocol. Faster aspart was titrated from randomisation (week 0) and onwards, twice weekly to reach the glycaemic target of pre-prandial and bedtime PG between 4.0-6.0 mmol/L (71 - 108 mg/dL) in a treat-to-target fashion.
- NovoRapid: Participants received insulin aspart (NovoRapid®/NovoLog®: basal-bolus regimen) with or without metformin for 16 weeks. Before the treatment period was a 12-week run-in period in which the investigator optimised basal insulin dose. Insulin degludec dose was adjusted weekly by the investigator in the run-in period based on the mean of three pre-breakfast SMPG values measured on the last two days prior to and on the day of contact. If one of the SMPG values were below target (< 4.0 mmol/L or 71 mg/dL) then the insulin degludec dose was adjusted according to the titration guideline specified in the protocol. NovoRapid was titrated from randomisation (week 0) and onwards, twice weekly to reach the glycaemic target of pre-prandial and bedtime PG between 4.0-6.0 mmol/L (71 - 108 mg/dL) in a treat-to-target fashion.
Period: Overall Study
Arm/Group | Faster Aspart | NovoRapid
Started | 546 | 545
Full Analysis Set | 546 | 545
Safety Analysis Set | 544 | 544
Completed | 531 | 531
Not Completed | 15 | 14
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawal by Subject | 11 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Faster Aspart | NovoRapid | Total
Number analyzed (Participants) | 546 | 545 | 1091
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.6 (8.6) | 62.1 (8.8) | 62.3 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 281 | 256 | 537
  Male | 265 | 289 | 554
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 487 | 487 | 974
    Asian | 43 | 31 | 74
    Black or African American | 14 | 19 | 33
    Native Hawaiian or Other Pacific Islander | 2 | 5 | 7
    Other | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Ethnicity
  Participants
    Not Hispanic or Latino | 485 | 488 | 973
    Hispanic Latino | 61 | 57 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline (week 0) in glycosylated haemoglobin (HbA1c) was evaluated at week 16. The endpoint was evaluated based on data from the in-trial observation period. In-trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Groups:
- NovoRapid: Participants received Insulin aspart (NovoRapid®/NovoLog®: basal-bolus regimen) along with insulin degludec (basal-bolus regimen) with or without metformin for 16 weeks. Before the treatment period was a 12-week run-in period in which the investigator optimised basal insulin dose. Insulin degludec dose was adjusted weekly by the investigator in the run-in period based on the mean of three pre-breakfast SMPG values measured on the last two days prior to and on the day of contact. If one of the SMPG values were below target (< 4.0 mmol/L or 71 mg/dL) then the insulin degludec dose was adjusted according to the titration guideline specified in the protocol. NovoRapid was titrated from randomisation (week 0) and onwards, twice weekly to reach the glycaemic target of pre-prandial and bedtime PG between 4.0-6.0 mmol/L (71 - 108 mg/dL) in a treat-to-target fashion.
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 539
Percentage of HbA1c | -0.15 (0.62) | -0.09 (0.60)
Statistical Analysis 1: Comparison: Faster Aspart vs NovoRapid; Change from baseline in HbA1c was analysed using an analysis of variance model after multiple imputation assuming treatment according to randomisation. The model included treatment, region and metformin use at baseline (Yes/No) as factors, and baseline HbA1c as a covariate; Test type: Non-Inferiority — The upper limit of the 95% confidence interval for the difference between faster aspart and NovoRapid was compared to a non-inferiority margin of 0.4%. If it was below or equal to 0.4% non-inferiority was considered established and effect demonstrated; p = 0.310, ANOVA; Treatment difference = -0.04, 95% CI 2-sided [-0.11 to 0.03] — Faster aspart-NovoRapid

2. Secondary Outcome: Change From Baseline in 1-hour PPG Increment
Description: Change from baseline (week 0) in 1-hour postprandial glucose (PPG) increment was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 519 | 523
mmol/L | -0.43 (2.45) | 0.08 (2.65)

3. Secondary Outcome: Change From Baseline in 1,5-anhydroglucitol
Description: Change from baseline (week 0) in 1,5-anhydroglucitol was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 534 | 531
mmol/L | 1.38 (3.10) | 0.89 (3.31)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG)
Description: Change from baseline (week 0) in fasting plasma glucose was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 533 | 530
mmol/L | 0.56 (2.38) | 0.68 (2.40)

5. Secondary Outcome: Participants Who Achieved HbA1c <7.0% (53 mmol/L) (Yes/No)
Description: Number of participants reaching HbA1c <7.0% (53 mmol/L) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: 16 weeks after randomisation
Population: Overall number of participants analyzed = full analysis set (FAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
Participants
  Yes | 271 | 282
  No | 275 | 263

6. Secondary Outcome: Participants Who Achieved HbA1c <7.0% (53 mmol/L) Without Severe Hypoglycaemia Episodes (Yes/No)
Description: Number of participants reaching HbA1c <7.0% (53 mmol/L) without severe hypoglycaemia episodes was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: 16 weeks after randomisation
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
Participants
  Yes | 265 | 278
  No | 281 | 267

7. Secondary Outcome: Change From Baseline (Week 0) in 30-minute, 1-hour, 2-hour, 3-hour and 4-hour Postprandial Glucose (PPG [Meal Test])
Description: Change from baseline (week 0) in 30-minute, 1-hour, 2-hour, 3-hour and 4-hour postprandial glucose (PPG [meal test]) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact. Meal test: The subjects were given a carbohydrate-rich standardised liquid meal immediately after bolus (faster aspart or NovoRapid) infusion in the morning of the meal test. The subjects were to consume the meal as quickly as possible (within 12 minutes) and blood samples were drawn after 30 minutes, 1, 2, 3 and 4 hours from the start of the meal.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
mmol/L
  30-min: number analyzed (Participants) | 519 | 522
  30-min | 0.31 (2.90) | 0.55 (2.80)
  1-hour: number analyzed (Participants) | 521 | 526
  1-hour | 0.03 (3.30) | 0.68 (3.23)
  2-hour: number analyzed (Participants) | 519 | 524
  2-hour | 0.08 (3.96) | 0.61 (3.48)
  3-hour: number analyzed (Participants) | 518 | 519
  3-hour | 0.30 (3.85) | 0.89 (3.72)
  4-hour: number analyzed (Participants) | 514 | 519
  4-hour | 0.51 (3.47) | 0.75 (3.51)

8. Secondary Outcome: Change From Baseline (Week 0) in 30-minute, 1-hour, 2-hour, 3-hour and 4-hour PPG Increment (Meal Test)
Description: Change from baseline (week 0) in 30-minute, 1-hour, 2-hour, 3-hour and 4-hour PPG increment (meal test) was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact. Meal test: The subjects were given a carbohydrate-rich standardised liquid meal immediately after bolus (faster aspart or NovoRapid) infusion in the morning of the meal test. The subjects were to consume the meal as quickly as possible (within 12 minutes) and blood samples were drawn after 30 minutes, 1, 2, 3 and 4 hours from the start of the meal. PPG incremental value for each time point was derived as PPG value at that time point minus the preprandial glucose value.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
mmol/L
  30-min: number analyzed (Participants) | 518 | 519
  30-min | -0.13 (1.85) | -0.05 (1.95)
  1-hour: number analyzed (Participants) | 519 | 523
  1-hour | -0.43 (2.45) | 0.08 (2.65)
  2-hour: number analyzed (Participants) | 517 | 521
  2-hour | -0.37 (3.25) | 0.001 (3.13)
  3-hour: number analyzed (Participants) | 516 | 516
  3-hour | -0.15 (3.23) | 0.28 (3.54)
  4-hour: number analyzed (Participants) | 513 | 516
  4-hour | 0.04 (3.00) | 0.15 (3.45)

9. Secondary Outcome: Change From Baseline in Mean of the 7-9-7 Point Self-measured Plasma Glucose (SMPG) Profile
Description: Change from baseline (week 0) in mean of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. 7-9-7 point SMPG was measured at the following mentioned time points: 1) Before breakfast, 2) 60 mins after the start of Breakfast, 3) Before lunch, 4) 60 mins after the start of lunch, 5) Before main evening meal, 6) 60 mins after the start of main evening meal, 7) At bedtime, 8) At 4 AM, 9) Before breakfast.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 454 | 464
mmol/L | -0.56 (1.66) | -0.50 (1.61)

10. Secondary Outcome: Change From Baseline of the 7-9-7 Point SMPG Profile: PPG (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in PPG (breakfast, lunch, main evening meal and mean over all meals) of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
mmol/L
  Breakfast: number analyzed (Participants) | 447 | 462
  Breakfast | -0.38 (2.53) | -0.28 (2.44)
  Lunch: number analyzed (Participants) | 453 | 462
  Lunch | -0.78 (2.48) | -0.58 (2.68)
  Main evening meal: number analyzed (Participants) | 447 | 459
  Main evening meal | -1.04 (2.67) | -0.71 (2.50)
  All meals: number analyzed (Participants) | 440 | 457
  All meals | -0.75 (1.89) | -0.52 (1.91)

11. Secondary Outcome: Change From Baseline of the 7-9-7 Point SMPG Profile: PPG Increment (Mean, Breakfast, Lunch and Main Evening Meal)
Description: Change from baseline (week 0) in PPG increment (breakfast, lunch, main evening meal and mean over all meals) of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. PPG increment based on the 7-9-7-point profiles were derived separately for PG measurements made at 1 hour after main meals (breakfast, lunch and main evening meal). PPG incremental value for each time point was derived as PPG value at that time point minus the preprandial glucose value. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
mmol/L
  Breakfast: number analyzed (Participants) | 447 | 461
  Breakfast | -0.56 (2.23) | -0.42 (2.17)
  Lunch: number analyzed (Participants) | 453 | 460
  Lunch | -0.38 (2.69) | -0.23 (2.46)
  Main evening meal: number analyzed (Participants) | 444 | 459
  Main evening meal | -0.44 (2.61) | -0.10 (2.28)
  All meals: number analyzed (Participants) | 438 | 455
  All meals | -0.48 (1.55) | -0.23 (1.42)

12. Secondary Outcome: Change From Baseline of the 7-9-7 Point SMPG Profile: Fluctuation in 7-9-7 Point Profile
Description: Fluctuation in 7-point SMPG profile was the average absolute difference from the mean of the SMPG profile. Reported results are fluctuation in the 7-9-7 point SMPG profile from baseline (week 0) after 16 weeks of randomisation (i.e., week 16). The results are presented as ratio to baseline. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 454 | 464
Ratio | 0.82 (48.32) | 0.85 (55.06)

13. Secondary Outcome: Change From Baseline of the 7-9-7 Point SMPG Profile: Nocturnal SMPG Measurements
Description: Change from baseline (week 0) in nocturnal SMPG measurements was assessed by considering the differences between PG values available at bedtime, at 4 AM and the before breakfast value the following day: (4 AM PG value minus at bedtime PG value), (before breakfast PG value minus at bedtime PG value) and (before breakfast PG value minus 4 AM PG value). Change from baseline in nocturnal increments in SMPG measurements of the 7-9-7 point SMPG profile was evaluated after 16 weeks of randomisation and presented during three different time intervals as follows: 1) 04:00 to breakfast, 2) bedtime to 04:00, and 3) bedtime to breakfast. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
mmol/L
  Bedtime to 04:00: number analyzed (Participants) | 343 | 347
  Bedtime to 04:00 | 0.70 (4.09) | 0.29 (4.09)
  Bedtime to breakfast: number analyzed (Participants) | 419 | 438
  Bedtime to breakfast | 1.30 (4.25) | 0.90 (3.99)
  04:00 to breakfast: number analyzed (Participants) | 351 | 355
  04:00 to breakfast | 0.66 (2.76) | 0.75 (2.87)

14. Secondary Outcome: Participants Who Achieved Overall PPG (1 Hour) <7.8 mmol/L (140 mg/dL) (Yes/No)
Description: Participants reaching overall PPG (1 hour) ≤7.8 mmol/L [140 mg/dL] was evaluated after 16 weeks of randomisation. Participants without a postprandial glucose measurement at week 16 were considered not to have achieved HbA1c target at week 16. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: 16 weeks after randomisation
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
Participants
  Yes | 186 | 192
  No | 360 | 353

15. Secondary Outcome: Participants Who Achieved Overall PPG <7.8 mmol/L (140 mg/dL) Without Severe Hypoglycaemia Episodes (Yes/No)
Description: Participants reaching overall PPG (1 hour) ≤7.8 mmol/L [140 mg/dL] without severe hypoglycaemia episodes was evaluated after 16 weeks of randomisation. Participants without a postprandial glucose measurement at week 16 were considered not to have achieved HbA1c target at week 16. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: 16 weeks after randomisation
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
Participants
  Yes | 182 | 190
  No | 364 | 355

16. Secondary Outcome: Total Bolus Insulin Dose: in Units/Day
Description: Total bolus insulin dose (Units/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: 16 weeks from randomisation
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 542
Units/day | 54.72 (35.82) | 53.38 (35.35)

17. Secondary Outcome: Total Bolus Insulin Dose: in Units/kg/Day
Description: Total bolus insulin dose (Units/kg/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: 16 weeks from randomisation
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 542
Units/kg/day | 0.57 (0.33) | 0.55 (0.34)

18. Secondary Outcome: Total Basal Insulin Dose: in Units/Day
Description: Total basal insulin dose (Units/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: 16 weeks from randomisation
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units/day
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 542
Units/day | 63.76 (35.21) | 62.25 (36.03)

19. Secondary Outcome: Total Basal Insulin Dose: in Units/kg/Day
Description: Total basal insulin dose (Units/kg/day) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: 16 weeks from randomisation
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 542
Units/kg/day | 0.66 (0.32) | 0.64 (0.32)

20. Secondary Outcome: Individual Meal Insulin Dose: in Units
Description: Individual meal time bolus insulin dose (Units) for breakast, lunch and main evening meal was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: 16 weeks from randomisation
Population: Overall number of participants analyzed = safety analysis set (SAS) which comprised all randomised participants. Number Analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Units
  Breakfast: number analyzed (Participants) | 544 | 543
  Breakfast | 16.27 (12.04) | 15.52 (11.38)
  Lunch: number analyzed (Participants) | 544 | 543
  Lunch | 18.51 (12.09) | 17.96 (11.73)
  Daily main evening meal: number analyzed (Participants) | 544 | 542
  Daily main evening meal | 19.88 (13.46) | 19.85 (14.47)

21. Secondary Outcome: Individual Meal Insulin Dose: in Units/kg
Description: Individual meal time bolus insulin dose (Units/kg) for breakast, lunch and main evening meal was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: 16 weeks from randomisation
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units/kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Units/kg
  Breakfast: number analyzed (Participants) | 544 | 543
  Breakfast | 0.17 (0.12) | 0.16 (0.11)
  Lunch: number analyzed (Participants) | 544 | 543
  Lunch | 0.19 (0.11) | 0.19 (0.12)
  Daily main evening meal: number analyzed (Participants) | 544 | 542
  Daily main evening meal | 0.21 (0.13) | 0.20 (0.14)

22. Secondary Outcome: Change From Baseline in Lipids-lipoproteins Profile (Total Cholesterol, High Density Lipoproteins, Low Density Lipoproteins) - Ratio to Baseline
Description: Reported results are lipids-lipoproteins (total cholesterol, high density lipoproteins, low density lipoproteins) values are given as ratio to baseline (week 0) after 16 weeks. The results are based on the last in-trial value, which included the last available measurement in the in-trial period. In trial observation period was from date of randomisation and until last trial-related participant-site contact.
Time Frame: Week 0, week 16
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 546 | 545
Ratio
  Total cholesterol: number analyzed (Participants) | 542 | 537
  Total cholesterol | 1.01 (15.98) | 1.00 (17.09)
  High density lipoproteins: number analyzed (Participants) | 542 | 537
  High density lipoproteins | 0.97 (14.47) | 0.98 (17.57)
  Low density lipoproteins: number analyzed (Participants) | 542 | 537
  Low density lipoproteins | 0.99 (25.36) | 0.99 (40.51)

23. Secondary Outcome: Number of Treatment Emergent Adverse Events
Description: Number of treatment emergent adverse events were recorded from week 0 to week 16. The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Number; unit: Events
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Events | 667 | 643

24. Secondary Outcome: Number of Treatment Emergent Injection Site Reactions
Description: Number of treatment emergent injection site reactions were recorded from week 0 to week 16. The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Number; unit: Number of injection site reactions
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of injection site reactions | 3 | 1

25. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes (Hypos) According to the American Diabetes Association (ADA) and Novo Nordisk (NN) Definition: Overall
Description: ADA classification of hypos:
  1. Severe: Requiring assistance of another person to actively administer carbohydrate/glucagon/take other corrective actions. PG levels may not be available during an event, but neurological recovery following return of PG to normal is considered sufficient evidence that event was induced by a low PG level.
  2. Documented symptomatic: PG ≤3.9 mmol/L with symptoms.
  3. Asymptomatic: PG ≤3.9 mmol/L without symptoms.
  4. Probable symptomatic: No measurement with symptoms.
  5. Pseudo: PG >3.9 mmol/L with symptoms.
  6. Unclassifiable.
  NN classification of hypos:
  1. BG confirmed: PG <3.1 mmol/L with/without symptoms.
  2. Severe or BG confirmed symptomatic: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with symptoms.
  3. Severe or BG confirmed: Severe as per ADA and BG confirmed by PG <3.1 mmol/L with/without symptoms.
  4. Unclassifiable. Not able to self treat-unclassifiable: Not able to self treat but not classifiable as severe hypoglycaemia.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 18 | 14
  ADA: Documented symptomatic | 5038 | 6165
  ADA: Asymptomatic | 3761 | 3681
  ADA: Probable symptomatic | 68 | 68
  ADA: Pseudo | 145 | 75
  ADA: Unclassifiable | 3 | 3
  NN: BG confirmed | 2209 | 2735
  NN: Severe or BG confirmed symptomatic | 1490 | 2055
  NN: Severe or BG confirmed | 2227 | 2749
  NN: Unclassifiable | 6806 | 7257
  Not able to selftreat - unclassifiable | 0 | 0

26. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Daytime Hypoglycaemic Episodes (06:00-00:00 - Inclusive)
Description: Number of treatment emergent day time hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 06:00 and 00:00 (both included). The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 16 | 12
  ADA: Documented symptomatic | 4703 | 5700
  ADA: Asymptomatic | 3617 | 3484
  ADA: Probable symptomatic | 62 | 64
  ADA: Pseudo | 141 | 66
  ADA: Unclassifiable | 3 | 3
  NN: BG confirmed | 2016 | 2442
  NN: Severe or BG confirmed symptomatic | 1333 | 1814
  NN: Severe or BG confirmed | 2032 | 2454
  NN: Unclassifiable | 6510 | 6875
  Not able to selftreat - unclassifiable | 0 | 0

27. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Nocturnal Hypoglycaemic Episodes (00:01-05:59 - Inclusive)
Description: Number of treatment emergent nocturnal hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 00:01 and 05:59 (both included). The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 2 | 2
  ADA: Documented symptomatic | 335 | 465
  ADA: Asymptomatic | 144 | 197
  ADA: Probable symptomatic | 6 | 4
  ADA: Pseudo | 4 | 9
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 193 | 293
  NN: Severe or BG confirmed symptomatic | 157 | 241
  NN: Severe or BG confirmed | 195 | 295
  NN: Unclassifiable | 296 | 382
  Not able to selftreat - unclassifiable | 0 | 0

28. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Hypoglycaemic Episodes During First 1 Hour After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated during the first 1 hour after start of the meal. The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 2 | 0
  ADA: Documented symptomatic | 149 | 148
  ADA: Asymptomatic | 87 | 80
  ADA: Probable symptomatic | 11 | 8
  ADA: Pseudo | 2 | 4
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 72 | 65
  NN: Severe or BG confirmed symptomatic | 48 | 50
  NN: Severe or BG confirmed | 74 | 65
  NN: Unclassifiable | 177 | 175
  Not able to selftreat - unclassifiable | 0 | 0

29. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Hypoglycaemic Episodes During First 2 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated during the first 2 hours after start of the meal. The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 2 | 1
  ADA: Documented symptomatic | 465 | 446
  ADA: Asymptomatic | 201 | 159
  ADA: Probable symptomatic | 16 | 11
  ADA: Pseudo | 10 | 7
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 233 | 246
  NN: Severe or BG confirmed symptomatic | 181 | 212
  NN: Severe or BG confirmed | 235 | 247
  NN: Unclassifiable | 459 | 377
  Not able to selftreat - unclassifiable | 0 | 0

30. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and Novo Nordisk Definition: Hypoglycaemic Episodes During First 4 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated during the first 4 hours after start of the meal. The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 6 | 9
  ADA: Documented symptomatic | 1627 | 1882
  ADA: Asymptomatic | 852 | 744
  ADA: Probable symptomatic | 37 | 27
  ADA: Pseudo | 55 | 26
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 762 | 965
  NN: Severe or BG confirmed symptomatic | 557 | 820
  NN: Severe or BG confirmed | 768 | 974
  NN: Unclassifiable | 1809 | 1714
  Not able to selftreat - unclassifiable | 0 | 0

31. Secondary Outcome: Number of Treatment Emergent Hypoglycaemic Episodes According to the American Diabetes Association and NN Definition: Hypoglycaemic Episodes Occurring Between 2 to 4 Hours After Start of the Meal
Description: Number of treatment emergent hypoglycaemic episodes according to the ADA and NN definitions were evaluated between 2 to 4 hours after start of the meal. The results are based on the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Weeks 0-16
Population: as for outcome 20
Measure: Number; unit: Number of hypoglycaemic episodes
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Number of hypoglycaemic episodes
  ADA: Severe | 4 | 8
  ADA: Documented symptomatic | 1162 | 1436
  ADA: Asymptomatic | 651 | 585
  ADA: Probable symptomatic | 21 | 16
  ADA: Pseudo | 45 | 19
  ADA: Unclassifiable | 0 | 0
  NN: BG confirmed | 529 | 719
  NN: Severe or BG confirmed symptomatic | 376 | 608
  NN: Severe or BG confirmed | 533 | 727
  NN: Unclassifiable | 1350 | 1337
  Not able to selftreat - unclassifiable | 0 | 0

32. Secondary Outcome: Change From Baseline in Physical Examination
Description: Participants with physical examination findings, normal, abnormal NCS (non- clinically significant) and abnormal CS (clinically significant) at baseline (week 0) and week 16 presented. Results are based on the data from the on-treatment observation period, which was the time period from when a participant was randomised until the final scheduled visit, including any period after initiation of rescue medication and/or premature discontinuation of trial product. Results are presented for the following examinations: 1) Cardiovascular system 2) Central & Peripheral nervous system 3) Gastrointestinal system incl. mouth 4) Head, ears, eyes, nose, throat and neck 5) Musculoskeletal system 6) Respiratory system 7) Skin
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Participants
  Cardiovascular system (week 0): Normal | 459 | 460
  Cardiovascular system (week 0): Abnormal NCS | 79 | 79
  Cardiovascular system (week 0): Abnormal CS | 6 | 5
  Cardiovascular system (week 16): number analyzed (Participants) | 525 | 533
  Cardiovascular system (week 16): Normal | 448 | 457
  Cardiovascular system (week 16): Abnormal NCS | 71 | 72
  Cardiovascular system (week 16): Abnormal CS | 6 | 4
  Central and Peripheral nervous sys. (week 0): Normal | 398 | 404
  Central and Peripheral nervous sys. (week 0): Abnormal NCS | 133 | 127
  Central and Peripheral nervous sys. (week 0): Abnormal CS | 13 | 13
  Central and Peripheral nervous sys. (week 16): number analyzed (Participants) | 525 | 533
  Central and Peripheral nervous sys. (week 16): Normal | 383 | 400
  Central and Peripheral nervous sys. (week 16): Abnormal NCS | 128 | 122
  Central and Peripheral nervous sys. (week 16): Abnormal CS | 14 | 11
  Gastrointestinal sys. including mouth (Week 0): Normal | 491 | 485
  Gastrointestinal sys. including mouth (Week 0): Abnormal NCS | 53 | 59
  Gastrointestinal sys. including mouth (Week 0): Abnormal CS | 0 | 0
  Gastrointestinal sys. including mouth (week 16): number analyzed (Participants) | 525 | 533
  Gastrointestinal sys. including mouth (week 16): Normal | 480 | 476
  Gastrointestinal sys. including mouth (week 16): Abnormal NCS | 45 | 57
  Gastrointestinal sys. including mouth (week 16): Abnormal CS | 0 | 0
  Head, ears, eyes, nose, throat, neck (week 0): Normal | 498 | 492
  Head, ears, eyes, nose, throat, neck (week 0): Abnormal NCS | 43 | 48
  Head, ears, eyes, nose, throat, neck (week 0): Abnormal CS | 3 | 4
  Head, ears, eyes, nose, throat, neck (week 16): number analyzed (Participants) | 525 | 533
  Head, ears, eyes, nose, throat, neck (week 16): Normal | 485 | 483
  Head, ears, eyes, nose, throat, neck (week 16): Abnormal NCS | 40 | 49
  Head, ears, eyes, nose, throat, neck (week 16): Abnormal CS | 0 | 1
  Musculoskeletal system (week 0): Normal | 504 | 496
  Musculoskeletal system (week 0): Abnormal NCS | 36 | 42
  Musculoskeletal system (week 0): Abnormal CS | 4 | 6
  Musculoskeletal system (week 16): number analyzed (Participants) | 525 | 533
  Musculoskeletal system (week 16): Normal | 489 | 494
  Musculoskeletal system (week 16): Abnormal NCS | 32 | 33
  Musculoskeletal system (week 16): Abnormal CS | 4 | 6
  Respiratory system (week 0): Normal | 535 | 534
  Respiratory system (week 0): Abnormal NCS | 9 | 9
  Respiratory system (week 0): Abnormal CS | 0 | 1
  Respiratory system (week 16): number analyzed (Participants) | 525 | 533
  Respiratory system (week 16): Normal | 520 | 517
  Respiratory system (week 16): Abnormal NCS | 5 | 14
  Respiratory system (week 16): Abnormal CS | 0 | 2
  Skin (week 0): Normal | 438 | 429
  Skin (week 0): Abnormal NCS | 96 | 108
  Skin (week 0): Abnormal CS | 10 | 7
  Skin (week 16): number analyzed (Participants) | 525 | 533
  Skin (week 16): Normal | 418 | 430
  Skin (week 16): Abnormal NCS | 98 | 98
  Skin (week 16): Abnormal CS | 9 | 5

33. Secondary Outcome: Change From Baseline in Vital Signs: Systolic and Diastolic Blood Presure
Description: Change in vital signs - systolic and diastolic blood pressure from baseline (week 0) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 525 | 533
mmHg
  Systolic blood pressure | 0.4 (14.0) | -1.2 (14.8)
  Diastolic blood pressure | -0.4 (8.9) | -0.7 (8.9)

34. Secondary Outcome: Change From Baseline in Vital Signs: Pulse
Description: Change in vital signs - pulse from baseline (week 0) was evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Beats per min
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 525 | 533
Beats per min | 0.5 (9.0) | 0.03 (8.9)

35. Secondary Outcome: Change From Baseline in Electrocardiogram (ECG)
Description: Changes in electrocardiogram (ECG) from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Participants
  Week 0: Normal | 287 | 270
  Week 0: Abnormal NCS | 252 | 264
  Week 0: Abnormal CS | 5 | 10
  Week 16: number analyzed (Participants) | 525 | 533
  Week 16: Normal | 274 | 272
  Week 16: Abnormal NCS | 245 | 253
  Week 16: Abnormal CS | 6 | 8

36. Secondary Outcome: Change From Baseline in Fundoscopy/Fundus Photography
Description: Changes in fundoscopy/fundus photography from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: as for outcome 20
Measure: Count of Participants; unit: Participants
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 544 | 544
Participants
  Left eye (week 0): number analyzed (Participants) | 544 | 543
  Left eye (week 0): Normal | 225 | 219
  Left eye (week 0): Abnormal NCS | 287 | 297
  Left eye (week 0): Abnormal CS | 32 | 27
  Left eye (week 16): number analyzed (Participants) | 514 | 516
  Left eye (week 16): Normal | 205 | 198
  Left eye (week 16): Abnormal NCS | 278 | 288
  Left eye (week 16): Abnormal CS | 31 | 30
  Right eye (week 0): Normal | 224 | 217
  Right eye (week 0): Abnormal NCS | 288 | 300
  Right eye (week 0): Abnormal CS | 32 | 27
  Right eye (week 16): number analyzed (Participants) | 514 | 517
  Right eye (week 16): Normal | 208 | 194
  Right eye (week 16): Abnormal NCS | 276 | 297
  Right eye (week 16): Abnormal CS | 30 | 26

37. Secondary Outcome: Change From Baseline in Haematology - Haematocrit
Description: Changes in haematology - haematocrit from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
Percentage | 0.48 (2.47) | 0.35 (2.47)

38. Secondary Outcome: Change From Baseline in Haematology - Haemoglobin
Description: Changes in haematology - haemoglobin from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
mmol/L | -0.02 (0.47) | -0.04 (0.43)

39. Secondary Outcome: Change From Baseline in Haematology - Leukocytes
Description: Changes in haematology - leukocytes from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 leukocytes/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
10^9 leukocytes/L | 0.01 (1.60) | -0.01 (1.35)

40. Secondary Outcome: Change From Baseline in Haematology - Thrombocytes
Description: Changes in haematology - thrombocytes from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^9 thrombocytes/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 531 | 533
10^9 thrombocytes/L | -0.9 (37.1) | -1.3 (38.7)

41. Secondary Outcome: Change From Baseline in Haematology - Erythrocytes
Description: Changes in haematology - erythrocytes from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: 10^12 erythrocytes/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
10^12 erythrocytes/L | -0.02 (0.28) | -0.04 (0.27)

42. Secondary Outcome: Change From Baseline in Biochemistry - Alanine Aminotransferase (ALT)
Description: Changes in biochemistry - alanine aminotransferase from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
U/L | -0.1 (9.4) | 3.1 (65.4)

43. Secondary Outcome: Change From Baseline in Biochemistry - Alkaline Phosphatase
Description: Changes in biochemistry - alkaline phosphatase from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
U/L | 2.9 (22.6) | 2.2 (18.3)

44. Secondary Outcome: Change From Baseline in Biochemistry - Aspartate Aminotransferase (AST)
Description: Changes in biochemistry - aspratate aminotransferase from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
U/L | -0.2 (7.9) | 2.2 (45.7)

45. Secondary Outcome: Change From Baseline in Biochemistry - Albumin
Description: Changes in biochemistry - albumin from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
g/dL | 0.02 (0.25) | 0.01 (0.26)

46. Secondary Outcome: Change From Baseline in Biochemistry - Creatinine
Description: Changes in biochemistry - creatinine from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
umol/L | 0.1 (11.1) | 1.5 (13.2)

47. Secondary Outcome: Change From Baseline in Biochemistry - Potassium
Description: Changes in biochemistry - potassium from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
mmol/L | -0.001 (0.50) | 0.02 (0.43)

48. Secondary Outcome: Change From Baseline in Biochemistry - Sodium
Description: Changes in biochemistry - sodium from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
mmol/L | -0.6 (2.6) | -0.7 (2.8)

49. Secondary Outcome: Change From Baseline in Biochemistry - Total Bilirubin
Description: Changes in biochemistry - total bilirubin from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 531 | 536
umol/L | 0.1 (2.7) | 0.1 (3.0)

50. Secondary Outcome: Change From Baseline in Biochemistry - Total Protein
Description: Changes in biochemistry - total protein from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 532 | 536
g/dL | -0.01 (0.35) | -0.02 (0.36)

51. Secondary Outcome: Change From Baseline in Body Weight
Description: Changes in body weight from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 522 | 530
kg | 1.19 (2.95) | 1.12 (4.01)

52. Secondary Outcome: Change From Baseline in Body Mass Index (BMI)
Description: Change in the body mass index (BMI) from baseline (week 0) were evaluated after 16 weeks of randomisation. The results are based on the last on-treatment value, which included the last available measurement in the on-treatment period. On-treatment period started from date of first dose of randomised NovoRapid/faster aspart and to 7 days after day of last dose or day before initiation of ancillary treatment.
Time Frame: Week 0, week 16
Population: Overall number of participants analyzed = number of participants with available data.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Faster Aspart | NovoRapid
Number analyzed (Participants) | 522 | 530
kg/m^2 | 0.43 (1.04) | 0.40 (1.40)

ADVERSE EVENTS:
Time Frame: Week 0 to Week 16 + 7 days. All reported adverse events (AEs) are treatment emergent (i.e., TEAE).
Description: All presented AEs are TEAEs. A TEAE was defined as an event that had onset date on or after the first day of exposure to trial product and no later than 7 days after the last day of trial product administration. Results are based on the SAS which included all participants receiving at least one dose of randomised treatment.
Arm/Group | Faster Aspart | NovoRapid
All-Cause Mortality (participants affected / at risk) | 2/544 | 1/544
Serious Adverse Events (participants affected / at risk) | 38/544 | 40/544
Other Adverse Events (participants affected / at risk) | 32/544 | 33/544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (N=544) | NovoRapid (N=544)
Accidental overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 2 (2) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Aortic aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Aortic valve replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Arteriosclerosis coronary artery (Cardiac disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Bile duct obstruction (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac stress test abnormal (Investigations) | 1 (1) | 0 (0)
Carpal tunnel decompression (Surgical and medical procedures) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 2 (2)
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 1 (1) | 0 (0)
Device malfunction (Product Issues) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 0 (0) | 2 (2)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 4 (4) | 3 (3)
Hypoglycaemic unconsciousness (Nervous system disorders) | 3 (3) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 1 (2)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Obstructive pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Orchitis (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rapid eye movements sleep abnormal (Psychiatric disorders) | 1 (1) | 0 (0)
Rehabilitation therapy (Surgical and medical procedures) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Subclavian vein occlusion (Vascular disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 2 (2) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Varicose ulceration (Vascular disorders) | 0 (0) | 1 (1)
Vascular parkinsonism (Nervous system disorders) | 1 (1) | 0 (0)
Vitrectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 1 (1) | 0 (0)
Wrong product administered (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Faster Aspart (N=544) | NovoRapid (N=544)
Nasopharyngitis (Infections and infestations) | 32 (35) | 33 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more scientific publications may be prepared collaboratively by the investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for up to 60 days to protect intellectual property.

DOCUMENTS (2):
  • Study Protocol (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03268005/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT03268005/SAP_001.pdf